CLINICAL TRIAL: NCT03661190
Title: Impact of Short-term Intensive Online Grammatical Reasoning Training on Cognition and Function in Adults Over 50: An Online Randomised Controlled Trial
Brief Title: Online Grammatical Reasoning Training for Older Adults
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); King's College London (Other); Wesnes Cognition Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 216941
Record Dates: First submitted 2018-07-30; First posted 2018-09-07 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grammatical Reasoning (Other): This group will complete a short-term Intensive Grammatical Reasoning cognitive task delivered online by Wesnes Cognition Ltd (START). Participants will be encouraged to complete the START training once a day for six-weeks.
  Interventions: Other: Grammatical Reasoning
- Control - Card Pairs (Other): The control group will complete a basic picture-matching task that will provide the same level of engagement, but without the learning effects.
  Interventions: Other: Card Pairs

INTERVENTIONS:
Other: Grammatical Reasoning — START measures the ability to determine the relationships among different shape combinations which are assigned to grammatical statements about them which can be either correct or incorrect. It is a measure of attention, working memory and executive control.
  Other Names: START
  Arms: Grammatical Reasoning
Other: Card Pairs — A basic picture-matching task.
  Arms: Control - Card Pairs

SUMMARY:
The START study will investigate the impact of playing a Grammatical Reasoning brain training task on overall brain function (cognition) and day-to-day function in people over 50.

The study builds on existing work that has shown very promising results with brain training approaches in older adults. There is good evidence that playing brain training games leads to improvements in brain functions including memory and reasoning. There is also a suggestion that regular involvement in brain training games might help reduce the risk of cognitive decline and dementia later in life. It appears that reasoning, or problem-solving, is particularly important as it is one of the first abilities to decline with age. This study will use this evidence to target reasoning in a specific brain training task. It will also explore the potential role of genetic factors in how people perform in the task.

The study will compare the impact of a Grammatical Reasoning Task (START) with a control task consisting of simple picture-matching. Over 7000 participants will be randomly allocated to either START or the control and will be asked to play the task as often as they wish for a period of six weeks. Both tasks will be delivered entirely online so people will access the study from home on their computers. This will be achieved through our dedicated online research platform, PROTECT, which hosts a cohort of over 20,000 older adults who have provided DNA samples as part of a longitudinal study.

This study will measure the impact of the training on cognition and Instrumental Activities of Daily Living. Assessments will be completed online at baseline, two/six weeks and six months. Overall, this study aims to generate exciting new data about how brain training could be included in guidance on healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50
* Access to a computer with a keyboard and the internet
* Participant registered on the PROTECT study

Exclusion Criteria:

* Diagnosis of dementia

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7240 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
A composite measure of cognitive function | Participants will be directed to complete these measures at baseline, two/ six weeks and six months
  The primary outcome measure will be a composite measure of cognitive function, created through a combined score of each of the measures described below. The individual measures will be included as discrete secondary outcome measures. All outcome measures will be completed online. They are sensitive to change in cognition, and validated for use in older adults to detect early changes in cognition.

SECONDARY OUTCOMES:
Executive function | Baseline, two weeks, six weeks and 6 months
  Measured by a test of visual attention, the Trail making B, which is a validated measure for use in this population.
Executive function | Baseline, two weeks, six weeks and 6 months
  Measured by a test of task-switching, the Switching Stroop Test, which is a validated measure for use in this population.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through the Baddeley Logical Reasoning Task (letter sequence)11 - part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Digit Vigilance test as part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Simple and Choice Reaction time test as part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Spatial Working Memory test as part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Numeric Working Memory test as part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Pattern Separation test as part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Word Recall (delayed and immediate) test as part of the Wesnes Cognition Ltd CogTrackTM system.
Cognitive function | Baseline, two weeks, six weeks and 6 months
  Measured through a Word Recognition test as part of the Wesnes Cognition Ltd CogTrackTM system.
Verbal Learning | Baseline, two weeks, six weeks and 6 months
  Measured through the validated Paired Associate Learning measure, which is highly sensitive to change in cognition and has been used to predict conversion to Alzheimer's Disease in people with cognitive impairment.
Instrumental Activities of Daily Living (IADL) | Baseline, two weeks, six weeks and 6 months
  Measured by the modified Instrumental Activities of Daily Living measure which is validated for use in this population, and has been successfully used to show change in IADL in previous online brain training studies.
Use of cognitive training | 6 months
  Participants will complete a brief question regarding their use of cognitive training (computer games, crosswords, Sudoku etc) and the regularity of use

CONTACTS AND LOCATIONS:
Overall Officials: Anne Corbett, BSc MRes PhD, Principal Investigator — University of Exeter Medical School
Locations (1):
- University of Exeter Medical School, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie results in a publication or for secondary data analysis purposes.